CLINICAL TRIAL: NCT03363802
Title: Assessment of Pubertal Growth Spurt in Growing Egyptian Females Using Modified Middle Phalanx of The Middle Finger Stages and Its Correlation With Development Stage of Mandibular Second Molar in Al Sharkia Governorate
Brief Title: Assessment of Pubertal Growth Spurt in Growing Girls Using Middle Phalynx Finger and Correlate With Mandibular Second Molar
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Magdy, Principal Investigator,Ms candidate, Cairo University
Other Study IDs: CEBC-CU-2017-12-01
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Growth Alteration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Assessment of Pubertal Growth Spurt in Growing Egyptian Females Using Modified Middle Phalanx of The Middle Finger Stages and Its Correlation With Development Stage of Mandibular Second Molar

DETAILED DESCRIPTION:
The sample will be selected randomly from different schools in the government.

* Digital periapical radiograph for the middle finger for each participants will be taken using Digital x-ray portable machine.
* Radiographical images will be stored in a digital sensor to be transferred to computer then we asses growth spurt in girls and correlate it with devlopemt stage of mandibular second molar

ELIGIBILITY:
Inclusion Criteria:

* Egyptian citizen

Exclusion Criteria:

* Systemic disease and syndromes
* Severe crowding

Ages: 9 Years to 14 Years | Sex: Female
Age Groups: Child
Study Population: Egyptian females between 9-14 years old to be sure that they are within or around the circumpubertal period.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2018-02-10 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of the time of pubertal growth spurt in growing Egyptian | 3month
  Taking xray of middle phalynx finger and then asses age of growth spurt through stages of middle phalynx finger

SECONDARY OUTCOMES:
females. Assessment the correlation between the modified middle phalanx of the middle finger and development stage of mandibular second molar | 3month
  By taking xray mandibular second molar then make correlation between stages of both to estimate age for pubertal growth spurt for females

CONTACTS AND LOCATIONS:
Locations (1):
- Schools, Zagazig, Sharkia Governorate, Egypt